CLINICAL TRIAL: NCT06421896
Title: Exploring the Motivational Enhancement Therapy's Impact on Motivation, Resilience, Anxiety Reduction, and COPD Outcomes in Geriatric Patient
Brief Title: Motivational Enhancement Therapy's Impact on d COPD Outcomes in Geriatric Patient
Acronym: METgeriatri
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 85-a
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group: geriatric who receive motivational Enhancement Therapy (Experimental): COPD geriatric patients who receive motivational Enhancement Therapy
  Interventions: Behavioral: motivational Enhancement Therapy
- non- experimental group (No Intervention): COPD geriatric patients who don't receive motivational Enhancement Therapy

INTERVENTIONS:
Behavioral: motivational Enhancement Therapy — Motivational Enhancement Therapy (MET) is a systematic intervention that focuses on eliciting and strengthening a person's intrinsic motivation to change. MET is rooted in motivational interviewing principles, emphasizing empathy, autonomy, and the evocation of the patient's own motivations for change. The therapy typically involves several sessions where therapists help patients identify personal goals, explore ambivalence towards change, and develop actionable plans to achieve their desired outcomes.
  Arms: experimental group: geriatric who receive motivational Enhancement Therapy

SUMMARY:
Motivational Enhancement Therapy (MET) is a systematic intervention that focuses on eliciting and strengthening a person's intrinsic motivation to change. MET is rooted in motivational interviewing principles, emphasizing empathy, autonomy, and the evocation of the patient's own motivations for change. The therapy typically involves several sessions where therapists help patients identify personal goals, explore ambivalence towards change, and develop actionable plans to achieve their desired outcomes.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of morbidity and mortality worldwide, particularly among the elderly. Managing COPD effectively in geriatric patients requires addressing not only the physiological aspects of the disease but also the psychological and motivational factors that can influence treatment adherence and overall well-being. Motivational Enhancement Therapy (MET) is a counseling approach designed to help individuals enhance their motivation to change and engage in healthier behaviors. This study explores the impact of MET on motivation, resilience, anxiety reduction, and COPD outcomes in geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* more than 60 years

Exclusion Criteria:

* more than 80 years

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
COPD geriatric patients who entered motivational Enhancement Therapy will demonstrate a higher score in resilience scale ( ( total score range from 15 to 75, a higher score of more than 50)than those who not entered | three months
  primary objective

SECONDARY OUTCOMES:
OPD geriatric patients who entered motivational Therapy will demonstrate a lower score in anxiety inventory ( total score range from 10 to 50, a lower score of more than 20)than those who not entered | three months
  secondary

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No